CLINICAL TRIAL: NCT04983251
Title: Women's Health Awareness Community Resiliency, Environmental Action and Collaborations for Health (REACH) Equity
Brief Title: Women s Health Awareness Community Resiliency, Environmental Action and Collaborations for Health (REACH) Equity
Status: Recruiting | Type: Observational
Sponsor: National Institute of Environmental Health Sciences (NIEHS) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 10000441; 000441-E
Record Dates: First submitted 2021-07-29; First posted 2021-07-30 (Actual); Last update posted 2025-12-10 (Actual); Status verified 2025-12-08

CONDITIONS: Mental Health
Keywords: Disparities; Vaccination; COVID-19; Natural History
MeSH Terms: conditions — Psychological Well-Being; COVID-19

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- U4 Women: Women in under-served, under-studied, under-represented, and under-reported (U4) populations.

SUMMARY:
Background:

Inequalities in COVID-19 infection, hospitalization, and death in under-studied, under-represented, and under-reported groups of people are severe. A growing number of studies have assessed the impact of individual risk factors. But few studies have assessed which factors are the greatest drivers of COVID-19 disparities from a wider perspective.

Objective:

To understand the long-term impacts of COVID-19 on minority women and their families to assist in developing community-based programs to help in recovery.

Eligibility:

Healthy people aged 18 and older who reside in North Carolina.

Design:

Participants will take a 45-minute online survey. The survey will cover their demographics, community, health, lifestyle, household, and environment.

Participants may choose to have tests. They may visit the Clinical Research Unit. They may also have a home visit for these tests. In some cases, they may mail samples to the study team in prepaid envelopes.

Participants may take an optional 15 minute survey about their reproductive history.

Participants may give a blood sample.

Participants may give a urine sample. They will fill out a log and return with their sample.

Participants may give saliva samples.

Participants may give toenail samples from each toe.

Participants may give dust samples. They will be given 8 alcohol swabs. Two will be for testing. They will be asked to swipe a total of 3 door frames. Each door frame should be in a different room of the house.

Participants may be given silicone wristbands to wear for 1 week. This is to measure their exposure to air pollutants.

Participants may be contacted in the future for follow-up. They may be contacted by phone, email, or letter.

DETAILED DESCRIPTION:
Study Description:

This is a cross-sectional population-based survey designed within a syndemic framework to characterize the impacts of the COVID-19 pandemic on women in under-served, under-studied, under-represented, and under-reported (U4) populations. We hypothesize that U4 women are experiencing and will have experienced a worsening of mental, physical, and socio-economic status as a result of the COVID-19 pandemic and that pre-pandemic indicators of U4 status and related exposures will be associated with adverse mental, physical, and SES effects of the COVID-19 pandemic. The study ultimately seeks to collect baseline data for a long-term follow-up study of U4 women, as well as identify high impact targets for public health interventions to build resiliency in U4 communities.

Objectives:

Primary Objectives:

1. Characterize the mental, physical, and socio-economic effects of the COVID-19 pandemic on women in under-served, under-studied, under-represented, and under-reported (U4) populations within a syndemic framework.
2. Determine whether there was a worsening of mental, physical, and socio-economic status before, during, and following the COVID-19 pandemic.
3. Characterize the biological, behavioral, environmental, sociocultural, and structural impacts of the COVID-19 pandemic on reproductive risk factors among U4 women.

Secondary Objectives:

1. Quantify cross-sectional associations between retrospective pre-pandemic indicators of U4 status and related exposures (i.e., urban vs. rural; pre-existing physical and mental health disparities; risk factors for maternal mortality; experiences of racism; social factors, and environmental, occupational, and housing exposures) with adverse mental, physical, and SES effects of the COVID-19 pandemic.
2. Characterize the direct and indirect experiences of U4 women with SARS-CoV-2 infection.
3. Identify opportunities for interventions to address maternal mortality in U4 women in the context of an ongoing global pandemic of COVID-19.

Tertiary/Exploratory Objectives:

1. Assess the association between geospatial indicators of exposure and pandemic impacts, including proximity to point sources of environmental pollution, area-level model and monitor-estimated air pollution concentrations, availability of community amenities, and neighborhood structure.
2. Collect baseline data for a future longitudinal cohort study on long-term health impacts of exposure to SARS-CoV-2 (COVID-19) and pandemic experiences among U4 women, as well as to identify risk and protective factors modifying these impacts for developing appropriate interventions for recovery in this population.
3. Pool data with ongoing COVID-19 observational studies to:

   (a) generalize pandemic impacts across multiple U4 populations using pooled meta-analysis; and (b) to understand how U4 status interacts with environmental, health, and social risk factors to produce disparities in pandemic-associated impacts by comparing U4 and non-U4 populations.
4. Understand the distribution and characteristics of exploratory cardiovascular biomarkers among U4 women of reproductive age and their relation to COVID-19 impacts, including SARS-CoV-2 infection and associations with a range of biological, behavioral, environmental, sociocultural, and structural factors impacted by the COVID-19 pandemic that affect pregnancy-related and pregnancy-associated morbidity and mortality.

Endpoints:

Primary. Characterization of mental health, physical health and socioeconomic impacts during and following the pandemic.

Secondary. Primary endpoints plus direct and indirect experiences with SARS-CoV-2 infection.

Tertiary/Exploratory.

1. Geospatial analyses

   1. Direct and indirect experiences with SARS-CoV-2 infection described above.
   2. Worsening of primary endpoints described above.
2. Longitudinal baseline

   1. History of chronic illness
   2. Interest in clinical research participation and acceptable methods
   3. Biological specimens (i.e., urinary cortisol; blood for SARS-CoV-2 antibody testing, cytokine profiling, reproductive endpoints; and blood and saliva for DNA methylation microarrays, toenail clippings for exposure)
   4. Personal exposure (i.e., home dust assays, personal exposure monitoring (wristband), toenail samples).
   5. First time point for repeated longitudinal stress and mental health assessments.
3. Meta-analysis

   1. Environmental, health, and social risk factors
   2. Pandemic-associated impacts

ELIGIBILITY:
* INCLUSION CRITERIA:

In order to be eligible to participate in this study, an individual must meet all of the following criteria:

1. Females who are African American or Black, Hispanic or Latino, American Indian or Alaska Native, Asian American, Native Hawaiian or other Pacific Islander.
2. Aged 18 years or older.
3. Reside in North Carolina.
4. Be willing to provide photo ID
5. Able to read and understand English in order to complete surveys (questions validated in English) and logs.

EXCLUSION CRITERIA:

An individual who meets any of the following criteria will be excluded from participation in this study:

-Any condition that, in the investigator's opinion, places the participant at undue risk for complications associated with required study procedures.

Ages: 18 Years to 100 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Women will be recruited from a community-based sample in North Carolina following a recruitment plan developed in collaboration with Women's Health Awareness (WHA) partners.
Sampling Method: Non-Probability Sample
Enrollment: 700 (Estimated)
Dates: Start 2023-06-30 (Actual); Primary Completion 2026-09-30 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Characterize the mental, physical, and socio-economic effects | 2 years
  (1)Characterize the mental, physical, and socio-economic effects of the COVID-19 pandemic on women in under-studied, under-represented, and under-reported (U4) populations within a syndemic framework. (2) Determine whether there was a worsening of mental, physical, and socio-economic status before, during, and following the COVID-19 pandemic. (3) Characterize the biological, behavioral, environmental, sociocultural, and structural impacts of the COVID-19 pandemic on factors that affect reproductive risk factors among U4 women.

SECONDARY OUTCOMES:
Quantify cross-sectional associations between retrospective pre-pandemic indicators of U4 status and related exposures | 2 years
  (1) Quantify cross-sectional associations between retrospective pre-pandemic indicators of U4 status and related exposures (i.e., urban vs. rural; pre-existing physical and mental health disparities; risk factors for maternal mortality; experiences of racism; social factors, and environmental, occupational, and housing exposures) with adverse mental, physical, and SES effects of the COVID-19 pandemic. (2) Characterize the direct and indirect experiences of U4 women with SARS-CoV-2 infection. (3) Identify opportunities for interventions to address maternal mortality in U4 women in the context of an ongoing global pandemic of COVID-19.

CONTACTS AND LOCATIONS:
Overall Officials: Joan P Packenham, Ph.D., Principal Investigator — National Institute of Environmental Health Sciences (NIEHS)
Locations (1):
- NIEHS Clinical Research Unit (CRU), Research Triangle Park, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_000441-E.html